CLINICAL TRIAL: NCT05670652
Title: Assessment of the Occlusal Characteristics of the Primary Dentition Among Egyptian Pre-School Children
Brief Title: Assessment of the Occlusal Characteristics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Faisal Ali Jarallah Aljarallah, Principal investigator, Cairo University
Other Study IDs: ocopd
Record Dates: First submitted 2022-12-06; First posted 2023-01-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Tooth Development Disorder
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: clinical examination — Clinical examination with optimal (Lighting, using a disposable mouth mirror and a millimeter-ruler) will be performed, in addition to an upper and lower arch impression will be made and a study cast will be prepared.

SUMMARY:
The objective of this study is to assess the occlusal characteristics of primary dentition among Egyptian preschool children.

DETAILED DESCRIPTION:
This cross-sectional study was based on examination of the primary dentition of healthy preschool Egyptian children ,The objective of this study is to assess the occlusal characteristics of primary dentition among Egyptian preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian children.
* Children are medically free.
* Children with a complete set of primary dentition without any permanent teeth. -Teeth free of extensive caries which affect the mesio- distal and occluso- gingival dimension.

Exclusion Criteria:

* Children with developmental anomalies.
* Children with any oral habits.
* Children with cognition problems.
* Children with a history of an obvious alternative cause for malocclusion (e.g. trauma, syndromes).
* Participant's caregivers refuse to give consent.

Ages: 3 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: Egyptian children aged from 3-6 years old
Sampling Method: Non-Probability Sample
Enrollment: 362 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Primary molar relationship | Day 1
  Categorical (Flush terminal plane, mesial step, distal step)

SECONDARY OUTCOMES:
Primary canine relationship | Day 1
  Categorical (Class 1, Class 2, Class3)
Physiological spaces (Upper and lower) | Day 1
  Binary (Present/absent)
Primate spaces (Upper and lower) | Day 1
  Binary (Present/absent)
Crowding (upper and lower) | Day 1
  Binary (Present/absent)
Midline discrepancy | Day 1
  Binary (Present/absent)
Posterior Crossbite (unilateral/bilateral) | Day 1
  Binary (Present/absent)
Degree of overbite | Day 1
  Categorical (Normal, increased, edge to edge or anterior open bite)
Degree of overjet | Day 1
  Categorical (Normal, increased, edge to edge or anterior crossbite)

CONTACTS AND LOCATIONS:
Overall Officials: Sherine Badr Youness, prof dr, Study Director — Cairo University; Shereen Hassan El-Shamy, dr, Study Director — Cairo University

REFERENCES:
- [Background] Davidopoulou S, Arapostathis K, Berdouses ED, Kavvadia K, Oulis C. Occlusal features of 5-year-old Greek children: a cross-sectional national study. BMC Oral Health. 2022 Jul 9;22(1):281. doi: 10.1186/s12903-022-02303-1. PMID 35810281
- [Background] BY Badr, S. and H Yahfoufi, S. (2020) 'ASSESSMENT OF THE OCCLUSALCHARACTERISTICS OF THE PRIMARY DENTITION AMONG LEBANESE PRE-SCHOOL CHILDREN: A BASE LINE STUDY CROSS-SECTIONAL STUDY', BAU Journal-Health and Wellbeing, 2(2), p. 5.
- [Background] El-Attar, H., Salama, R. and Hussien, A. (2020) 'Prevalence of malocclusion and common occlusal traits among adolescent school children in Dakahliya, Egypt and Makkah, Saudi Arabia (A comparative study)', Egyptian Orthodontic Journal, 57(June 2020), pp. 1-9.